CLINICAL TRIAL: NCT04110431
Title: Comparison Between Left Bundle Branch Pacing and Biventricular Pacing for Cardiac Resynchronization Therapy in Heart Failure(LBBP-RESYNC)
Brief Title: Left Bundle Branch Pacing Versus Biventricular Pacing for Cardiac Resynchronization Therapy
Acronym: LBBP-RESYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FirstNanjingMU002
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Chronic Heart Failure
Keywords: cardiac resynchronization therapy; chronic heart failure; left bundle branch pacing; biventricular pacing
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBP group (Experimental): In this arm, An right artrial (RA) lead and an implantable cardioverter defibrillator (ICD) lead are conventionally implanted. A left bundle branch pacing(LBBP) lead is attempted to be placed. If LBBP failed, a left ventricular(LV) pacing lead is implanted instead.
  Interventions: Procedure: Left bundle branch pacing
- BivP group (Active Comparator): In this arm, an RA lead , an ICD lead and a LV pacing lead are placed. If the implantation of LV pacing lead is unsuccessful due to unavailable coronary sinus branches(venae cordis magna or venae cordis media is not recommended), capture above 3.5V/0.5ms or refractory phrenic nerve stimulation,a LBBP lead is placed instead.
  Interventions: Procedure: Biventricular pacing

INTERVENTIONS:
Procedure: Left bundle branch pacing — Successful LBBP was defined as (1) LBBP lead is located at 1.5-2cm from His-bundle towards right ventricular apex; (2) Paced QRS morphology of right bundle branch delay(CRBBD) in lead V1; (3) Stimulus to the peak of R wave in V5 and V6 QRS wave, which represents left ventricular activation time(Stim-LVAT), is less than 100ms and constant at high and low output pacing; (4) Unipolar pacing threshold<1.5V/0.5ms; (5) Recording P potential when narrow QRS escape rhythm or CRBBB escape rhythm(not essential).
  Arms: LBBP group
Procedure: Biventricular pacing — Implantation of a LV pacing lead is attempted using the standard-of-care technique first.
  Arms: BivP group

SUMMARY:
The present study will recruit 40 symptomatic heart failure patients with left ventricular ejection fraction (LVEF) below 35% and complete left bundle branch block(QRSd≥130 ms). Each patient was randomized to either left bundle branch pacing(LBBP) or biventricular pacing(BivP) and was followed up for at least 6 months. The objective is to compare the effects of LBBP and BivP on cardiac resynchronization in the treatment of heart failure by measurable clinical parameters.

DETAILED DESCRIPTION:
The traditional biventricular pacing (BivP) is an established treatment to corrected the cardiac dyssynchrony in heart failure patients with left bundle branch block(LBBB). It has been proved that BivP can improve clinical symptoms and reduce all-cause mortality in heart failure. However, BivP is subject to the variable coronary sinus(CS) anatomy and LV-pacing lead fail to be implanted in 5%-10% of patients due to the lack of appropriate target branch, high threshold or phrenic nerve stimulation. Almost 30%-40% of patients with successful implantation show no response. What's more, BivP just corrects the mechanical dyssynchrony caused by LBBB not corrects the LBBB. Recent studies have demonstrated that His bundle pacing (HBP) can correct LBBB, achieve physiological pacing and realize the cardiac resynchronization. But HBP has high technical requirements, lower sense value and higher threshold of correcting LBBB, which may be further increased in long-term follow-up.

The lastest research shows that pacing left ventricular septum using a transseptal approach can reduce left ventricular(LV) electrical dyssynchrony. Huang et al first confirmed that left bundle branch pacing(LBBP) can correct LBBB and improve cardiac function. LBBP has been reported to offer higher success rate with higher sense value and lower pacing thresholds compared with HBP. In chronic heart failure patients with LBBB that need cardiac resynchronization therapy(CRT), LBBP can achieve the similar electrical and mechanical resynchronization as well as HBP.

There is to date no randomized studies between LBBP and BivP in HFrEF patients with complete LBBB that need CRT. The purpose of this study is to compare the therapeutic effects of LBBP and conventional BivP on LV function and clinical endpoints in such patients. The present study will randomize 40 patients in two centres to LBBP or BivP. Baseline assessments including echocardiography parameters[left ventricular ejection fraction(LVEF ), left ventricular end-systolic volume(LVESV), left ventricular end-diastolic volume(LVEDV)], electrocardiogram(ECG), N-terminal pro B-type natriuretic peptide(NT-proBNP) level, New York Heart Association(NYHA) class, 6-minute walking distance(6MWD) and quality of life score(QOL) will be obtained. At the same time, the LBBP and BivP success rate, intraoperative and postoperative complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

1. LVEF≤35% as assessed by echocardiography and NYHA class II-IV despite optimal medical therapy for at lest 3 months；
2. Sinus rhythm, complete left bundle branch block (QRS duration ≥130ms)；
3. Between the ages of 18 and 80；
4. With informed consent signed.

Exclusion Criteria:

1. After mechanical tricuspid valve replacement；
2. Unstable angina, acute MI, CABG or PCI within the past 3 months;
3. Persistent atrial fibrillation without atrioventricular block, the expected percentage of ventricular pacing below 95%;
4. Enrollment in any other study；
5. A life expectancy of less than 12 months；
6. Pregnant or with child-bearing potential;
7. History of heart transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Echocardiography parameters(LVEF,LVESV and LVEDV) | Baseline; 6-month follow-up
  Changes in LVEF,LVESV and LVEDV between baseline and follow-up

SECONDARY OUTCOMES:
Paced QRS duration | Postoperative day 1; 1-month,3-month and 6-month follow-upP
  Paced QRS duration is evaluated postoperative day 1 and 1 months, 3 months and 6 months after implantation.
Changes in concentration of NT-proBNP in blood between baseline and follow-up | Baseline; 1-month,3-month and 6-month follow-up
  Blood test is performed at each time frame to determine the concentration of NT-proBNP(unit: pg/mL)
Changes in New York Heart Association Heart Function Classification between baseline and follow-up | Baseline; 1-month,3-month and 6-month follow-up
  The higher the classification, the more severe the heart failure symptoms(four levels: I, II, III and IV)
Changes in 6-minute Walk Distance between baseline and follow-up | Baseline; 1-month,3-month and 6-month follow-up
  Distance that a participant walk within 6 minutes
Change in Quality Of Life Questionnaire score between baseline and follow-up | Baseline; 1-month,3-month and 6-month follow-up
  Reflect the effect of heart failure on quality of life, and higher scores represent a worse outcome
Incidence of clinical adverse events | 6-month follow-up
  Including date and number of all-cause mortality, heart failure hospitalization, cardiovascular hospitalization and malignant ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Zou, MD,Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Fu Wai Hospital, Beijing, China, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Background] Hou X, Qian Z, Wang Y, Qiu Y, Chen X, Jiang H, Jiang Z, Wu H, Zhao Z, Zhou W, Zou J. Feasibility and cardiac synchrony of permanent left bundle branch pacing through the interventricular septum. Europace. 2019 Nov 1;21(11):1694-1702. doi: 10.1093/europace/euz188. PMID 31322651
- [Background] Mafi-Rad M, Luermans JG, Blaauw Y, Janssen M, Crijns HJ, Prinzen FW, Vernooy K. Feasibility and Acute Hemodynamic Effect of Left Ventricular Septal Pacing by Transvenous Approach Through the Interventricular Septum. Circ Arrhythm Electrophysiol. 2016 Mar;9(3):e003344. doi: 10.1161/CIRCEP.115.003344. PMID 26888445
- [Derived] Wang Y, Zhu H, Hou X, Wang Z, Zou F, Qian Z, Wei Y, Wang X, Zhang L, Li X, Liu Z, Xue S, Qin C, Zeng J, Li H, Wu H, Ma H, Ellenbogen KA, Gold MR, Fan X, Zou J; LBBP-RESYNC Investigators. Randomized Trial of Left Bundle Branch vs Biventricular Pacing for Cardiac Resynchronization Therapy. J Am Coll Cardiol. 2022 Sep 27;80(13):1205-1216. doi: 10.1016/j.jacc.2022.07.019. PMID 36137670